CLINICAL TRIAL: NCT06818474
Title: Lanadelumab in Long-term Prophylaxis of Acquired Angioedema
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bernstein Clinical Research Center (Other)
Responsible Party: Principal Investigator, Jonathan A. Bernstein, MD, PI/ Owner, Bernstein Clinical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tak-02
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Angioedema
MeSH Terms: conditions — Angioedema | interventions — lanadelumab

STUDY DESIGN:
Intervention Model Description: all subjects will receive active treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- open-label administration (Other): all subjects receive open-label lanadelumab
  Interventions: Biological: Lanadelumab 300 mg

INTERVENTIONS:
Biological: Lanadelumab 300 mg — no other intervention

SUMMARY:
use of lanadelumab in patients with acquired angioedema

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of AAE with recurrent attacks without urticaria (decreased C1INH functional, quantitative levels, decreased C4 and decreased C1q levels, no family history of angioedema), presence of anti-C1INH antibody and/or paraproteinemia (e.g. monoclonal gammopathy of unknown significance)
* historical attack rate of >= on attack per month prior to starting tranexamic acid (TAA)

Exclusion Criteria:

* History of anaphylaxis or hypersensitivity to biologics
* History of major systemic disease not well controlled in opinion of the PI
* Women who are pregnant or breast feeding
* Concurrent participation in other clinical trials
* HAE Type 1 or 2 and normal complement HAE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 12 months
  Rate of investigator confirmed AAE attacks during study period, as measured by the ACT. AAE attack will be defined as a unique event during which the study subject will progress from no angioedema to symptoms of angioedema and no further angioedema for 24 hours after resolution of the event with rescu therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bernstein, MD, Principal Investigator — 5139314181
Locations (1):
- Bernstein Clinical Research Center, LLC, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided